CLINICAL TRIAL: NCT04058028
Title: A Phase 2b Dose Ranging Study to Evaluate the Efficacy and Safety of Rozibafusp Alfa (AMG 570) in Subjects With Active Systemic Lupus Erythematosus (SLE) With Inadequate Response to Standard of Care (SOC) Therapy
Brief Title: Efficacy and Safety of AMG 570 in Subjects With Active Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170588
Record Dates: First submitted 2019-07-30; First posted 2019-08-15 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Standard of Care therapies; Oral Corticosteroids; Inmunosuppressants; Immunomodulators; Systemic Lupus Erythematosus; B cell Activating Factor (BAFF); Inducible T cell costimulator ligand (ICOSL)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — rozibafusp alfa

STUDY DESIGN:
Intervention Model Description: This is a Bayesian adaptive phase 2b, multi-center, double-blind, randomized, placebo-controlled, 52-week, dose-ranging study in subjects with active SLE and inadequate response to SOC therapies including OCS, immunosuppressants, and immunomodulators. Subjects will be randomized to receive placebo or 1 of 3 doses of Rozibafusp Alfa with the last dose at week 50. Treatment will be administered every 2 weeks (Q2W). All subjects will be required to complete a 16-week follow-up period after the 52-week treatment period.
  The first interim analysis (IA) will be executed after the first 40 enrolled subjects have had the opportunity to complete the week 24 assessment. Additional IAs may be executed after approximately every 32 newly enrolled subjects have had the opportunity to complete the week 24 assessment. The last IA will occur when all subjects have had the opportunity to complete the week 24 assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Rozibafusp Alfa, Dose A (Experimental): Investigational product solution in vial
  Interventions: Drug: Rozibafusp Alfa
- Rozibafusp Alfa, Dose B (Experimental): Investigational product solution in vial
  Interventions: Drug: Rozibafusp Alfa
- Rozibafusp Alfa, Dose C (Experimental): Investigational product solution in vial
  Interventions: Drug: Rozibafusp Alfa
- Placebo for Rozibafusp Alfa (Placebo Comparator): Placebo Investigational product solution in vial
  Interventions: Drug: Placebo for Rozibafusp Alfa

INTERVENTIONS:
Drug: Rozibafusp Alfa — Rozibafusp Alfa will be presented in 5 mL glass vial
  Arms: Rozibafusp Alfa, Dose A; Rozibafusp Alfa, Dose B; Rozibafusp Alfa, Dose C
Drug: Placebo for Rozibafusp Alfa — Placebo for Rozibafusp Alfa will be presented in 5 mL glass vial
  Arms: Placebo for Rozibafusp Alfa

SUMMARY:
The purpose of this study is to determine if Rozibafusp Alfa could be a useful therapeutic agent in the current treatment landscape where subjects with SLE have ongoing disease activity despite treatment with standard of care therapies.

DETAILED DESCRIPTION:
This is a Bayesian adaptive phase 2b, multi-center, double-blind, randomized, placebo-controlled, 52-week, dose-ranging study in subjects with active SLE and inadequate response to SOC therapies including oral corticosteroids (OCS), immunosuppressants and immunomodulators. Previous biologic use is allowed with an adequate washout period.

ELIGIBILITY:
Inclusion Criteria Screening Visit:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures.
* Age ≥ 18 years to ≤ 75 years at screening visit.
* Fulfills classification criteria for SLE according to the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for SLE (Aringer et al, 2019), with antinuclear antibody ≥ 1:80 by immunofluorescence on Hep-2 cells being present at screening.
* Hybrid SLEDAI score ≥ 6 points with a "Clinical" hSLEDAI score ≥ 4 points. The "Clinical" hSLEDAI is the hSLEDAI assessment score without the inclusion of points attributable to laboratory results, including urine or immunologic parameters.
* Additional protocol-specific rules are applied at screening and throughout the study, as follows:

  * Arthritis: Arthritis (at least 3 tender and swollen joints) must involve joints in the hands or wrists for the hSLEDAI scoring.
  * Alopecia: Subjects should have hair loss without scarring; should neither have alopecia areata nor androgenic alopecia; and should have a CLASI activity score for alopecia ≥ 2.
  * Oral ulcers: Ulcers location and appearance must be documented by the investigator.
  * Scleritis and Episcleritis: the presence of stable SLE-related scleritis and episcleritis must be documented by an ophthalmologist and other causes excluded.
  * Renal: subjects with urine protein/creatinine ratio < 3000 mg/g (or equivalent method) in a clear catch spot urine sample can enroll and be scored in the hSLEDAI, provided the subject has a clinical hSLEDAI ≥ 4 and did not receive induction treatment for nephritis within the last year.
  * Pleurisy and Pericarditis: symptoms of pleurisy and pericarditis must be accompanied by objective findings to be scored in the hSLEDAI.
* Unless there is a documented intolerance, subjects must be taking:

  * Only 1 of the following SLE treatments: anti-malarial (hydroxychloroquine, chloroquine, or quinacrine), azathioprine, methotrexate, leflunomide, mycophenolate mofetil/acid mycophenolic, or dapsone.

OR

• 2 of the above-mentioned SLE treatments in which 1 must be anti-malarial (hydroxychloroquine, chloroquine, or quinacrine).

* Treatment should be taken for ≥ 12 weeks prior to screening and must be a stable dose for ≥ 8 weeks prior to screening.
* For subjects taking OCS, dose must be ≤ 20 mg/day of prednisone or OCS equivalent, and the dose must be stable at baseline visit for ≥ 2 weeks prior to screening visit.

Exclusion Criteria Screening Visit

Subjects are excluded from the study if any of the following criteria apply:

Disease Related

* Urine protein creatinine ratio ≥ 3000 mg/g (or equivalent) at screening or induction therapy for lupus nephritis within 1 year prior to screening visit.
* Active CNS lupus within 1 year prior to screening including, but not limited to, aseptic meningitis, ataxia, CNS vasculitis, cranial neuropathy, demyelinating syndrome, optic neuritis, psychosis, seizures, or transverse myelitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (147):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Imaging Endpoints, Scottsdale, Arizona
  - Medvin Clinical Research, Covina, California
  - Southern California Permanente Medical Group, Fontana, California
  - University of California San Diego, La Jolla, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University Hospitals and Clinics, Palo Alto, California
  - TriWest Research Associates, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Centre for Rheumatology Immunology and Arthritis, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Lakes Research LLC, Miami Lakes, Florida
  - Heuer Medical Doctor Research LLC, Orlando, Florida
  - Southwest Florida Clinical Research Center, Tampa, Florida
  - AdventHealth Medical Group, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Clinic of Robert Hozman, MD - Clinical Investigational Specialists, Inc, Skokie, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland School of Medicine Division of Rheumatology, Baltimore, Maryland
  - Feinstein Institute for Medical Research, Manhasset, New York
  - New York University Langone Orthopedic Center, New York, New York
  - Hospital For Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - DJL Clinical Research PLLC, Charlotte, North Carolina
  - Arthritis and Rheumatology Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - The Oklahoma Center for Arthritis Therapy and Research Inc, Tulsa, Oklahoma
  - Penn State Milton South Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Articularis Healthcare Group Inc dba Low Country Rheumatology, Summerville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Regional Clinic Specialty Research, Austin, Texas
  - Trinity Universal Research Associates, Inc, Carrollton, Texas
  - Rheumatic Disease Clinical Research Center LLC, Houston, Texas
  - Southwest Rheumatology, Mesquite, Texas
- Argentina (8):
  - Dom Centro de Reumatologia, CABA, Buenos Aires
  - Fundacion Respirar - Centro Medico Dra De Salvo, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Instituto Medico de Alta Complejidad San Isidro, San Isidro, Buenos Aires
  - Hospital Militar Central - Cirujano Mayor Dr Cosme Argerich, Buenos Aires, Distrito Federal
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Clinical Mayo - Clinica Mayo de Urgencias Medicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - CER San Juan - Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
- Australia (2):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment Trimontium OOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment - Kaspela EOOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Medical Center Excelsior OOD, Sofia
  - Medical Center Academy EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Sveti Ivan Rilski EAD, Sofia
  - Medical Centre Synexus Sofia EOOD, Sofia
  - Medical Centre Synexus Sofia EOOD - Branch Stara Zagora, Stara Zagora
- Canada (3):
  - University of Calgary Cumming School of Medicine, Calgary, Alberta
  - Shared Health Inc. operating the Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Groupe de recherche en maladies osseuses Incorporated, Québec, Quebec
- Czechia (2):
  - Synexus Czech sro, Prague
  - Revmatologicky ustav, Prague
- France (9):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Pellegrin, Bordeaux
  - CHU Hôpital Côte de Nacre, Caen
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hopital Francois Mitterrand, Dijon
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Claude Huriez, Lille
  - Hopital Pitie-Salpetriere, Paris
  - Centre Hospitalier Universitaire de Reims - Hopital Robert Debre, Reims
  - Centre Hospitalier Universitaire de Strasbourg - Nouvel hopital civil, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Purpan, Toulouse
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
- Germany (2):
  - Johannes Gutenberg Universitaet Mainz, Bad Kreuznach
  - Universitätsklinikum Leipzig AöR, Leipzig
- Greece (4):
  - Laiko General Hospital, Athens
  - Attiko Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - General University Hospital of Patras Panagia i Voithia, Pátrai
- Tuen Mun Hospital, New Territories, Hong Kong
- Hungary (3):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Vita Verum Medical Bt, Székesfehérvár
- Italy (4):
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Policlinico Universitario Agostino Gemelli, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
- Japan (21):
  - National Hospital Organization Chibahigashi National Hospital, Chiba, Chiba
  - Juntendo University Urayasu Hospital, Urayasu-shi, Chiba
  - Hospital of the University of Occupational and Environmental Health Japan, Kitakyushu-shi, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - National University Corporation Tohoku University Tohoku University Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto-shi, Nagano
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - National Hospital Organization Nagasaki Medical Center, Omura-shi, Nagasaki
  - Sasebo Chuo Hospital, Sasebo-shi, Nagasaki
  - Kurashiki Medical Clinic, Kurashiki-shi, Okayama-ken
  - Okayama University Hospital, Okayama, Okayama-ken
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - St Lukes International Hospital, Chuo-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
- Mexico (6):
  - Centro Medico del Angel SC, Mexicali, Baja California Norte
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicalli, Baja California Norte
  - Morales Vargas Centro de Investigacion SC, León, Guanajuato
  - Centro Integral en Reumatologia SA de CV, Guadalajara, Jalisco
  - Centro Peninsular de Investigación Clínica, Mérida, Yucatán
  - Centro Mexicano de Desarrollo de Estudios Clinicos, Mexico City
- Poland (15):
  - Synexus Polska Spzoo, Gdansk
  - Synexus Polska Spzoo, Gdynia
  - Synexus Polska Spzoo, Katowice
  - Silmedic Spzoo, Katowice
  - Tomed Tomasz Miszalski-Jamka Centrum Medyczne, Krakow
  - Synexus Polska Spzoo, Lodz
  - Somed cr, Lodz
  - 1 Wojskowy Szpital Kliniczny z Poliklinika Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Lublin
  - Clinical Best Solutions Spolka z ograniczona odpowiedzialnoscia Spolka komandytowa, Lublin
  - Synexus Polska Spzoo, Poznan
  - Sanus Szpital Specjalistyczny Spzoo, Stalowa Wola
  - SOMED CR, Warsaw
  - Synexus Polska Spolka z ograniczona odpowiedzialnoscia, Warsaw
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Wroclaw
  - Synexus Polska Spzoo, Wroclaw
- Portugal (5):
  - Hospital Garcia de Orta, EPE, Almada
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - Centro Hospitalar Universitario de Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto EPE - Hospital de Santo Antonio, Porto
  - Centro Hospitalar Universtario de Sao Joao, EPE, Porto
- Russia (8):
  - Limited liability company Scientific Research Medical Complex Your Health, Kazan'
  - LLC Medical Center Maksimum Zdorovia, Kemerovo
  - LLC Medical center Revma Med, Kemerovo
  - FSBSI SRI of Rheumatology na V A Nasonova, Moscow
  - LLC Center of medicine Healthy family, Novosibirsk
  - LLC Center of general medicine, Novosibirsk
  - LLC Medical Sanitary Unit №157, Saint Petersburg
  - State Budget Medical Institution Sverdlovsk Regional Clinical Hospital N1, Yekaterinburg
- South Korea (4):
  - Keimyung University Dongsan Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ajou University Hospital, Suwon-si, Gyeonggi-do
- Spain (3):
  - Hospital Infanta Luisa, Seville, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Garces S, Karis E, Merrill JT, Askanase AD, Kalunian K, Mo M, Milmont CE. Improving resource utilisation in SLE drug development through innovative trial design. Lupus Sci Med. 2023 Jul;10(2):e000890. doi: 10.1136/lupus-2022-000890. PMID 37491104
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with active systemic lupus erythematosus (SLE) were recruited across 81 centers in Argentina, Bulgaria, Canada, Czech Republic, France, Germany, Greece, Hong Kong, Hungary, Italy, Japan, Mexico, Poland, Portugal, Russia, South Korea, Spain, and the United States from February 2020 to July 2023.
Pre-assignment Details: Response adaptive randomization was used to assign eligible participants to receive rozibafusp alfa at 70, 280, and 420 mg administered subcutaneously (SC) every 2 weeks (Q2W), or matching placebo. Randomization started with a 1:1:1:1 ratio and was subsequently adapted according to clinical efficacy.
Groups:
- Placebo: Participants received matching placebo for a maximum duration of 52 weeks.
- Rozibafusp Alfa 70mg: Participants received Rozibafusp Alfa 70mg SC Q2W for a maximum duration of 52 weeks.
- Rozibafusp Alfa 280mg: Participants received Rozibafusp Alfa 280mg SC Q2W for a maximum duration of 52 weeks.
- Rozibafusp Alfa 420mg: Participants received Rozibafusp Alfa 420mg SC Q2W for a maximum duration of 52 weeks.
Period: Overall Study
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Started | 62 | 58 | 36 | 88
Completed | 36 | 44 | 28 | 46
Not Completed | 26 | 14 | 8 | 42
Not completed — Withdrawal of Consent from Study | 12 | 8 | 6 | 7
Not completed — Decision by Sponsor | 13 | 4 | 1 | 35
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg | Total
Number analyzed (Participants) | 62 | 58 | 36 | 88 | 244
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (10.3) | 44.6 (12.3) | 42.2 (10.5) | 44.0 (10.5) | 43.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 33 | 82 | 228
  Male | 5 | 2 | 3 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 14 | 5 | 25 | 68
  Not Hispanic or Latino | 37 | 44 | 31 | 63 | 175
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 2 | 3
  Asian | 3 | 6 | 2 | 8 | 19
  Black (or African American) | 4 | 4 | 4 | 5 | 17
  Multiple | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 0 | 0
  White | 53 | 47 | 30 | 71 | 201
  Other | 2 | 0 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a SLE Responder Index (SRI-4) Response at Week 52
Description: SRI-4 response at Week 52 is defined as a ≥ 4-point decrease in the hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI) score, and no new British Isles Lupus Assessment Group (BILAG) 2004 A score, no greater than 1 new BILAG B domain scores compared with baseline, and a less than 0.3-point deterioration from baseline in Physician Global Assessment (PGA) (scale 0 to 3), and no use of more than protocol allowed therapies.
Time Frame: Week 52
Population: The FAS included all randomized participants. Only participants who had the opportunity to complete the visit by the date of the study termination decision being communicated to sites were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 43 | 51 | 35 | 48
Participants | 26 | 29 | 21 | 35

2. Secondary Outcome: Number of Participants With a SRI-4 Response at Week 24
Description: SRI-4 response at Week 24 is defined as a ≥ 4-point decrease in the hSLEDAI score, and no new BILAG 2004 A score, no greater than 1 new BILAG B domain scores compared with baseline, and a less than 0.3-point deterioration from baseline in PGA (scale 0 to 3), and no use of more than protocol allowed therapies.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 54 | 58 | 36 | 66
Participants | 33 | 30 | 20 | 46

3. Secondary Outcome: Number of Participants Who Achieved a BILAG Based Combined Lupus Assessment (BICLA) Response at Week 24
Description: The BICLA response is defined as:
  1. An improvement in baseline BILAG domain scores across all body systems with moderate (domain B) or severe disease activity (domain A)
  2. No new BILAG 2004 A domain score and no > 1 new BILAG 2004 B domain scores compared with baseline
  3. No worsening of the hSLEDAI score from baseline
  4. No ≥ 0.3-point deterioration from baseline in PGA
  5. No use of more than protocol-allowed therapies
  6. No disallowed changes in concomitant medications, mainly including increases in corticosteroids, immunosuppressants.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 54 | 58 | 36 | 66
Participants | 24 | 19 | 18 | 35

4. Secondary Outcome: Number of Participants Who Achieved a Lupus Low Disease Activity State (LLDAS) Response at Week 52
Description: LLDAS was defined as meeting all the following conditions:
  1. hSLEDAI ≤ 4, with no activity in major organ system (renal, central nervous system [CNS], cardiopulmonary, vasculitis, fever) and hemolytic anemia or gastrointestinal activity
  2. No new lupus disease activity as compared with the previous assessment
  3. PGA ≤ 1 (on a scale of 0 to 3)
  4. Current prednisone or equivalent dose of ≤ 7.5 mg/day
  5. Well-tolerated standard maintenance doses of immunosuppressive drugs and approved treatments, as allowed and specified in the protocol.
Time Frame: Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 43 | 51 | 35 | 48
Participants | 12 | 18 | 6 | 21

5. Secondary Outcome: Number of Participants Who Achieved a BICLA Response at Week 52
Description: as for outcome 3
Time Frame: Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 43 | 51 | 35 | 48
Participants | 21 | 20 | 15 | 29

6. Secondary Outcome: Number of Participants Achieving a SRI-4 Response With a Reduction of Oral Corticosteroids (OCS) to ≤ 7.5 mg/Day by Week 44 and Sustained Through Week 52 In Participants With a Baseline OCS Dose ≥ 10 mg/Day
Description: SRI-4 response is defined as a ≥ 4-point decrease in the hSLEDAI score, and no new BILAG 2004 A score, no greater than 1 new BILAG B domain scores compared with baseline, and a less than 0.3-point deterioration from baseline in PGA (scale 0 to 3), and no use of more than protocol allowed therapies. Participants also had to meet a reduction if OCS to ≤ 7.5 mg/day by Week 44 sustained through Week 52.
Time Frame: Up to Week 52
Population: The FAS included all randomized participants. Only participants who had a baseline OCS dose ≥ 10 mg/day and had the opportunity to complete Week 52 visit by the date of the study termination were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 27 | 16 | 19 | 25
Participants | 5 | 1 | 2 | 8

7. Secondary Outcome: Annualized Moderate and Severe Flare Rate Over 52 Weeks as Measured by Safety of Estrogens in Systemic Lupus Erythematosus National Assessment [SELENA] -Systemic Lupus Erythematosus Disease Activity Index [SLEDAI] Flare Index (SFI)
Description: The SFI, serves as a composite outcome measure incorporating the SELENA-SLEDAI score, and classifications of flares into mild, moderate, and severe, along with the PGA of disease activity. The SFI details specific clinical manifestations for each organ system and categorizes flares into mild, moderate, and severe based on treatment decisions. Moderate and severe flare: • Moderate: meeting criteria like SELENA-SLEDAI score change of 3 to 12 points, SLE symptom development, prednisone dose increase, non-steroidal anti-inflammatory drugs (NSAIDs)/hydrochloroquine addition, or PGA score increase by 1 to 2.5. • Severe: meeting criteria like SELENA-SLEDAI increase over 12 points, onset or worsening of severe symptoms, significant prednisone dose escalation, introduction of potent immunosuppressants, hospitalization, or PGA score reaching 2.5 or higher. Annualized flare rate was calculated as the number of flares divided by flare exposure time in days, multiplied by 365.25 for each Group.
Time Frame: Up to Week 52
Population: The FAS included all randomized participants.
Measure: Number; unit: Flares/year
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 62 | 58 | 36 | 88
Flares/year | 0.34 | 0.52 | 0.46 | 0.34

8. Secondary Outcome: Annualized Severe Flare Rate Over 52 Weeks as Measured by SFI
Description: The SFI, serves as a composite outcome measure incorporating the SELENA-SLEDAI score, and classifications of flares into mild, moderate, and severe, along with the PGA of disease activity. The SFI details specific clinical manifestations for each organ system and categorizes flares into mild, moderate, and severe based on treatment decisions. Severe flare: meeting criteria like SELENA-SLEDAI increase over 12 points, onset or worsening of severe symptoms, significant prednisone dose escalation, introduction of potent immunosuppressants, hospitalization, or PGA score reaching 2.5 or higher. The annualized flare rate was calculated as the number of flares divided by the flare exposure time in days, multiplied by 365.25 for each Group.
Time Frame: Up to Week 52
Population: The FAS included all randomized participants.
Measure: Number; unit: Flares/year
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 62 | 58 | 36 | 88
Flares/year | 0.21 | 0.24 | 0.30 | 0.16

9. Secondary Outcome: Annualized Flares Rate Over 52 Weeks as Measured by BILAG Score Designation of "Worse" or "New" Resulting in a B-Score In ≥ 2 Organs or an A-Score in ≥ 1 Organ
Description: The BILAG flare index was derived from BILAG 2004, as measured by BILAG score designation of 'worse' or 'new' resulting in a B score in >= 2 organs or an A score in >= 1 organ.
  The annualized flare rate was calculated as the number of flares divided by the flare exposure time in days, multiplied by 365.25 for each Group.
Time Frame: Up to Week 52
Population: The FAS included all randomized participants.
Measure: Number; unit: Flares/year
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 62 | 58 | 36 | 88
Flares/year | 0.13 | 0.22 | 0.30 | 0.31

10. Secondary Outcome: Number of Participants With ≥6 Tender and Swollen Joints in Hands and Wrists at Baseline Achieving ≥50% Improvement From Baseline at Weeks 12, 24, 36, and 52
Description: The tender and swollen joint count is a physical assessment where for each swollen and tender joint a score of 1 is assigned. Scores are then summed up to provide a total score for both swollen and tender joints. Higher total score indicate a severe disease activity and a lower score indicates a lees severe disease activity.
Time Frame: Week 12, 24, 36, and 52
Population: The FAS included all randomized participants. Only participants who had ≥ 6 tender and swollen joints involving hands and wrists at baseline and had opportunity to complete the visit by the date of the study termination were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 34 | 35 | 13 | 46
Participants
  Week 12 | 20 | 16 | 8 | 31
  Week 24: number analyzed (Participants) | 32 | 35 | 13 | 39
  Week 24 | 23 | 23 | 7 | 34
  Week 36: number analyzed (Participants) | 31 | 34 | 12 | 34
  Week 36 | 26 | 22 | 10 | 29
  Week 52: number analyzed (Participants) | 26 | 29 | 12 | 30
  Week 52 | 19 | 20 | 9 | 27

11. Secondary Outcome: Number of Participants With a Cutaneous Lupus Erythematosus Area and Severity Index (CLASI) Activity Score ≥8 at Baseline Achieving ≥50% Improvement From Baseline at Weeks 12, 24, 36, and 52
Description: The CLASI is an assessment tool consisting of two scores: one for disease activity and one for damage. Activity Score: Ranges from 0 to 70, and is assessed based on erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss, and non-scarring alopecia. Higher scores indicate more severe disease activity.
  Damage Score: Ranges from 0 to 56, and is evaluated through dyspigmentation and scarring, including scarring alopecia. Dyspigmentation that remains visible for more than 12 months is considered permanent, and its score is doubled. Higher scores indicate greater damage.
Time Frame: Week 12, 24, 36, and 52
Population: The FAS included all randomized participants. Only participants who had CLASI activity score ≥ 8 at baseline and had the opportunity to complete the visit by the date of the study termination were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 13 | 10 | 12 | 16
Participants
  Week 12 | 3 | 2 | 5 | 4
  Week 24: number analyzed (Participants) | 10 | 10 | 12 | 11
  Week 24 | 3 | 3 | 6 | 3
  Week 36: number analyzed (Participants) | 9 | 10 | 12 | 8
  Week 36 | 1 | 5 | 7 | 2
  Week 52: number analyzed (Participants) | 8 | 9 | 12 | 7
  Week 52 | 0 | 4 | 7 | 3

12. Secondary Outcome: Change From Baseline in Patient-Reported Outcome Measurement Information System Fatigue Short Form 7a Instrument (PROMIS-Fatigue SF7a) Score at Weeks 12, 24, 36, 44, and 52
Description: The PROMIS-Fatigue SF7a is a 7-item instrument that assesses the experience of fatigue as well as its impact on physical, mental and social activities. Each item is scored on a 5-point Likert scale, ranging from "1" (Never) to "5" (Always). The scores of all 7 items are summed up with a total raw score range of 7(low level of fatigue)-35(high level of fatigue). Raw scores are converted to a T-score ranging from 29.4(low level of fatigue)-83.2(high level of fatigue).
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 30 | 28 | 22 | 43
T-score
  Week 12 | -8.40 (9.61) | -6.89 (5.71) | -4.22 (8.45) | -8.01 (7.60)
  Week 24: number analyzed (Participants) | 27 | 25 | 14 | 31
  Week 24 | -6.48 (11.97) | -5.61 (8.54) | -5.86 (7.76) | -8.82 (6.02)
  Week 36: number analyzed (Participants) | 22 | 23 | 14 | 23
  Week 36 | -7.26 (8.26) | -7.12 (8.00) | -3.26 (7.64) | -8.73 (8.98)
  Week 44: number analyzed (Participants) | 22 | 24 | 17 | 23
  Week 44 | -4.44 (7.94) | -8.65 (9.75) | -4.47 (7.23) | -8.25 (10.38)
  Week 52: number analyzed (Participants) | 19 | 21 | 15 | 21
  Week 52 | -8.57 (8.36) | -10.22 (8.89) | -6.57 (7.25) | -7.88 (11.88)

13. Secondary Outcome: Change From Baseline in the Short Form 36 Version 2 (SF-36v2) Health Survey Physical Component Score at Weeks 12, 24, 36, 44 and 52
Description: The SF-36v2 (acute version) Health Survey consists of 36 items and serves as a patient-reported measure of health status. It assesses 8 domains of health-related quality of life: physical limitations, social limitations, role limitations due to physical health, bodily pain, mental health, role limitations due to emotional health, vitality, and general health perceptions. Each domain of the SF-36v2 produces a score ranging from 0 to 100, with higher scores indicating better health-related quality of life.
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 67
Score on a scale
  Week 12 | 4.612 (8.241) | 4.261 (7.609) | 4.013 (8.456) | 5.409 (6.207)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 50
  Week 24 | 6.055 (8.043) | 5.440 (8.807) | 4.570 (8.994) | 5.847 (6.971)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 44
  Week 36 | 6.652 (7.957) | 6.536 (9.646) | 5.360 (8.736) | 6.833 (9.467)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Week 44 | 4.881 (9.200) | 7.298 (9.903) | 3.508 (7.538) | 7.522 (9.735)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Week 52 | 7.235 (7.097) | 6.598 (9.452) | 5.056 (9.429) | 5.456 (9.151)

14. Secondary Outcome: Change From Baseline in the SF-36v2 Health Survey Mental Component Score at Weeks 12, 24, 36, 44 and 52
Description: as for outcome 13
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 67
Score on a scale
  Week 12 | 5.433 (10.477) | 1.941 (8.689) | 2.235 (11.754) | 4.965 (9.413)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 50
  Week 24 | 4.889 (10.772) | 1.123 (7.767) | 5.008 (8.063) | 5.786 (9.278)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 44
  Week 36 | 5.002 (9.405) | 1.407 (10.943) | 2.111 (11.263) | 6.531 (10.543)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Week 44 | 6.556 (12.984) | 3.208 (9.125) | 1.914 (9.247) | 5.903 (10.847)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Week 52 | 6.675 (12.074) | 3.778 (9.910) | 2.613 (10.841) | 7.186 (9.185)

15. Secondary Outcome: Change From Baseline in the SF-36v2 Health Survey Physical Functioning Domain Score at Weeks 12, 24, 36, 44 and 52
Description: as for outcome 13
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 68
Score on a scale
  Week 12 | 14.019 (25.397) | 11.383 (21.076) | 10.000 (22.966) | 12.595 (18.765)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 51
  Week 24 | 15.777 (23.930) | 13.043 (22.961) | 13.000 (24.657) | 14.048 (21.031)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 45
  Week 36 | 17.752 (22.417) | 15.640 (21.031) | 11.608 (23.533) | 16.142 (21.924)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 37
  Week 44 | 15.001 (24.582) | 17.222 (24.007) | 8.036 (19.924) | 17.200 (20.702)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 36
  Week 52 | 20.807 (21.138) | 15.416 (23.002) | 12.778 (22.632) | 16.568 (18.357)

16. Secondary Outcome: Change From Baseline in the SF-36v2 Health Survey Physical Role Domain Score at Weeks 12, 24, 36, 44 and 52
Description: as for outcome 13
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 67
Score on a scale
  Week 12 | 15.074 (25.378) | 7.979 (24.090) | 9.961 (21.701) | 13.713 (22.957)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 50
  Week 24 | 20.278 (28.240) | 10.190 (28.788) | 11.667 (19.609) | 16.625 (27.217)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 44
  Week 36 | 19.219 (24.160) | 12.660 (29.991) | 13.839 (23.653) | 19.886 (30.863)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Week 44 | 16.319 (28.554) | 18.924 (28.169) | 10.714 (22.876) | 20.313 (32.915)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Week 52 | 23.387 (22.475) | 17.708 (27.730) | 9.028 (23.852) | 14.464 (31.933)

17. Secondary Outcome: Change From Baseline in the SF-36v2 Health Survey Bodily Pain Domain Score at Weeks 12, 24, 36, 44 and 52
Description: as for outcome 13
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 67
Score on a scale
  Week 12 | 15.5 (25.7) | 12.0 (23.1) | 10.9 (21.5) | 18.4 (19.5)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 50
  Week 24 | 17.5 (26.7) | 14.4 (27.6) | 13.5 (24.6) | 18.3 (19.4)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 44
  Week 36 | 18.7 (23.2) | 15.9 (27.9) | 14.1 (24.0) | 22.1 (26.3)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Week 44 | 18.9 (23.9) | 19.2 (31.9) | 10.7 (20.5) | 26.0 (29.4)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Week 52 | 19.8 (22.5) | 16.7 (28.4) | 16.6 (23.0) | 21.8 (25.2)

18. Secondary Outcome: Change From Baseline in the SF-36v2 Health Survey General Health Domain Score at Weeks 12, 24, 36, 44 and 52
Description: as for outcome 13
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 68
Score on a scale
  Week 12 | 5.90 (14.71) | 5.85 (16.06) | 4.69 (14.87) | 9.97 (14.15)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 51
  Week 24 | 7.44 (15.97) | 6.98 (16.11) | 9.13 (14.83) | 11.75 (14.11)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 45
  Week 36 | 10.35 (16.43) | 10.15 (16.97) | 5.96 (16.28) | 11.40 (17.81)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 37
  Week 44 | 7.61 (19.32) | 11.81 (18.99) | 3.11 (16.92) | 11.76 (16.74)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 36
  Week 52 | 9.55 (21.62) | 12.54 (18.23) | 5.81 (19.60) | 9.58 (18.22)

19. Secondary Outcome: Change From Baseline in the SF-36v2 Health Survey Vitality Domain Score at Weeks 12, 24, 36, 44 and 52
Description: as for outcome 13
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 67
Score on a scale
  Week 12 | 10.662 (22.441) | 8.112 (18.054) | 8.594 (21.402) | 11.287 (20.361)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 50
  Week 24 | 10.556 (24.419) | 7.880 (15.780) | 12.083 (18.346) | 13.125 (18.482)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 44
  Week 36 | 11.094 (20.090) | 10.256 (19.102) | 8.036 (18.854) | 15.199 (22.083)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Week 44 | 7.465 (24.313) | 11.632 (19.489) | 5.804 (19.089) | 15.104 (21.670)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Week 52 | 12.903 (23.659) | 11.806 (20.199) | 8.796 (21.249) | 11.250 (21.693)

20. Secondary Outcome: Change From Baseline in the SF-36v2 Health Survey Social Role Functioning Domain Score at Weeks 12, 24, 36, 44 and 52
Description: as for outcome 13
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 67
Score on a scale
  Week 12 | 14.46 (22.83) | 8.24 (20.40) | 9.77 (24.54) | 15.11 (23.89)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 50
  Week 24 | 15.28 (26.23) | 7.88 (25.05) | 14.58 (19.72) | 15.25 (21.32)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 44
  Week 36 | 15.63 (25.28) | 7.05 (25.78) | 14.29 (23.00) | 19.60 (23.72)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Week 44 | 17.71 (27.61) | 8.68 (27.52) | 7.14 (22.16) | 14.24 (23.75)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Week 52 | 23.79 (25.07) | 10.42 (26.98) | 13.89 (23.34) | 17.50 (21.90)

21. Secondary Outcome: Change From Baseline in the SF-36v2 Health Survey Emotional Role Domain Score at Weeks 12, 24, 36, 44 and 52
Description: as for outcome 13
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 67
Score on a scale
  Week 12 | 13.888 (26.961) | 5.141 (26.384) | 2.083 (27.189) | 12.935 (27.382)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 50
  Week 24 | 13.888 (27.352) | 5.072 (23.339) | 11.111 (20.800) | 15.334 (28.540)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 44
  Week 36 | 15.208 (24.306) | 4.058 (21.364) | 6.250 (29.886) | 14.773 (29.742)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Week 44 | 20.139 (32.512) | 8.564 (21.314) | 7.441 (25.493) | 16.899 (30.045)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Week 52 | 18.011 (30.814) | 10.647 (25.008) | 6.481 (28.620) | 19.762 (23.491)

22. Secondary Outcome: Change From Baseline in the SF-36v2 Health Survey Mental Health Domain Score at Weeks 12, 24, 36, 44 and 52
Description: as for outcome 13
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 47 | 32 | 67
Score on a scale
  Week 12 | 10.7 (21.5) | 4.3 (16.2) | 6.4 (21.0) | 8.9 (17.1)
  Week 24: number analyzed (Participants) | 45 | 46 | 30 | 50
  Week 24 | 10.1 (22.7) | 2.7 (15.3) | 9.2 (15.1) | 10.6 (18.0)
  Week 36: number analyzed (Participants) | 40 | 39 | 28 | 44
  Week 36 | 10.0 (18.7) | 5.5 (21.8) | 3.0 (20.2) | 13.1 (19.3)
  Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Week 44 | 11.8 (24.3) | 10.3 (16.0) | 3.0 (16.1) | 12.5 (20.1)
  Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Week 52 | 12.3 (21.4) | 9.0 (19.0) | 4.6 (17.4) | 13.9 (18.3)

23. Secondary Outcome: Change From Baseline in Lupus Quality of Life Questionnaire (LupusQoL) Score at Weeks 12, 24, 36, 44, and 52
Description: The LupusQoL questionnaire consists of 8 domains: physical health, pain, planning, intimate relationships, burden to others, emotional health, body image, and fatigue. Each item in the questionnaire is scored on a 5 point scale and items within a given domain are summed and converted to a 0-100 scale. Each domain is scored 0-100 with higher scores representing better quality of life in the specific domain. Lower scores signify poorer quality of life within the domain.
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 46 | 32 | 67
Score on a scale
  Planning: Week 12 | 10.294 (23.368) | 11.594 (21.551) | 5.469 (23.817) | 12.438 (22.631)
  Planning: Week 24: number analyzed (Participants) | 45 | 45 | 30 | 50
  Planning: Week 24 | 10.185 (23.763) | 6.667 (29.226) | 9.722 (24.279) | 9.500 (23.988)
  Planning: Week 36: number analyzed (Participants) | 41 | 40 | 27 | 44
  Planning: Week 36 | 11.179 (21.214) | 9.583 (23.232) | 13.272 (21.836) | 14.773 (29.414)
  Planning: Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Planning: Week 44 | 9.491 (26.959) | 13.426 (20.919) | 9.821 (19.779) | 12.037 (27.418)
  Planning: Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Planning: Week 52 | 16.129 (19.357) | 8.565 (23.527) | 9.568 (24.428) | 12.381 (22.810)
  Physical Health: Week 12 | 9.498 (22.989) | 12.160 (15.607) | 8.398 (20.992) | 9.748 (16.541)
  Physical Health: Week 24: number analyzed (Participants) | 45 | 45 | 30 | 50
  Physical Health: Week 24 | 12.986 (24.461) | 14.097 (21.972) | 11.667 (18.856) | 11.063 (16.551)
  Physical Health: Week 36: number analyzed (Participants) | 41 | 40 | 27 | 44
  Physical Health: Week 36 | 12.729 (21.678) | 14.375 (22.610) | 13.542 (17.313) | 13.991 (21.264)
  Physical Health: Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Physical Health: Week 44 | 11.892 (25.253) | 16.753 (22.124) | 11.049 (15.625) | 12.760 (17.008)
  Physical Health: Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Physical Health: Week 52 | 18.448 (22.827) | 13.976 (19.799) | 8.449 (20.156) | 14.107 (18.847)
  Pain: Week 12 | 14.869 (27.199) | 14.493 (22.800) | 12.240 (26.939) | 14.552 (22.349)
  Pain: Week 24: number analyzed (Participants) | 45 | 45 | 30 | 50
  Pain: Week 24 | 16.296 (29.460) | 13.148 (22.647) | 15.556 (23.947) | 17.667 (20.800)
  Pain: Week 36: number analyzed (Participants) | 41 | 40 | 27 | 44
  Pain: Week 36 | 14.837 (26.972) | 13.125 (19.327) | 15.123 (23.912) | 18.939 (27.159)
  Pain: Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Pain: Week 44 | 14.815 (31.755) | 16.667 (23.905) | 11.905 (21.328) | 17.824 (24.893)
  Pain: Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Pain: Week 52 | 25.538 (23.367) | 14.352 (24.929) | 14.815 (28.898) | 19.524 (23.565)
  Intimate Relationship: Week 12: number analyzed (Participants) | 37 | 32 | 21 | 50
  Intimate Relationship: Week 12 | 6.76 (26.94) | 3.52 (24.64) | 0.60 (30.99) | 4.75 (20.81)
  Intimate Relationship: Week 24: number analyzed (Participants) | 29 | 32 | 18 | 34
  Intimate Relationship: Week 24 | 2.59 (24.86) | 5.47 (28.74) | 0.69 (20.77) | 6.25 (23.08)
  Intimate Relationship: Week 36: number analyzed (Participants) | 27 | 27 | 19 | 29
  Intimate Relationship: Week 36 | 4.63 (26.66) | 9.26 (27.21) | -2.63 (20.66) | 5.17 (23.27)
  Intimate Relationship: Week 44: number analyzed (Participants) | 25 | 25 | 19 | 26
  Intimate Relationship: Week 44 | 5.00 (31.46) | 8.00 (23.90) | -3.95 (21.67) | 9.13 (31.54)
  Intimate Relationship: Week 52: number analyzed (Participants) | 21 | 23 | 17 | 27
  Intimate Relationship: Week 52 | 11.90 (27.80) | 3.26 (23.30) | -1.47 (18.69) | 4.17 (19.61)
  Burden to Others: Week 12: number analyzed (Participants) | 51 | 26 | 32 | 67
  Burden to Others: Week 12 | 12.092 (22.068) | 5.072 (20.373) | 13.281 (30.590) | 9.577 (27.762)
  Burden to Others: Week 24: number analyzed (Participants) | 45 | 45 | 30 | 50
  Burden to Others: Week 24 | 10.556 (30.896) | 9.444 (27.328) | 15.000 (25.931) | 11.500 (27.914)
  Burden to Others: Week36: number analyzed (Participants) | 41 | 40 | 27 | 44
  Burden to Others: Week36 | 16.260 (27.320) | 11.042 (22.754) | 18.827 (28.457) | 13.447 (29.268)
  Burden to Others: Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Burden to Others: Week 44 | 14.120 (28.159) | 14.352 (23.955) | 15.476 (26.324) | 13.194 (26.902)
  Burden to Others: Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Burden to Others: Week 52 | 13.710 (27.348) | 8.333 (25.973) | 15.741 (30.865) | 17.143 (29.632)
  Emotional Health: Week 12 | 7.435 (23.940) | 4.529 (15.611) | 6.250 (21.997) | 9.142 (19.493)
  Emotional Health: Week 24: number analyzed (Participants) | 45 | 45 | 30 | 50
  Emotional Health: Week 24 | 8.056 (22.322) | 7.963 (19.337) | 7.778 (16.109) | 13.083 (22.096)
  Emotional Health: Week 36: number analyzed (Participants) | 41 | 40 | 27 | 44
  Emotional Health: Week 36 | 5.589 (19.557) | 3.958 (16.150) | 6.173 (20.359) | 13.920 (25.903)
  Emotional Health: Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Emotional Health: Week 44 | 6.134 (23.369) | 9.722 (15.685) | 7.292 (15.533) | 13.194 (23.853)
  Emotional Health: Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Emotional Health: Week 52 | 7.258 (23.545) | 6.134 (19.606) | 8.951 (20.888) | 14.167 (21.561)
  Body Image: Week 12 | 9.2 (24.4) | 3.7 (23.9) | 13.1 (31.7) | 10.1 (23.9)
  Body Image: Week 24: number analyzed (Participants) | 45 | 45 | 30 | 50
  Body Image: Week 24 | 5.9 (26.2) | -0.1 (24.9) | 0.2 (29.7) | 14.9 (26.4)
  Body Image: Week 36: number analyzed (Participants) | 41 | 40 | 27 | 44
  Body Image: Week 36 | 4.4 (25.0) | 3.8 (24.3) | 4.8 (27.7) | 11.1 (29.2)
  Body Image: Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Body Image: Week 44 | 11.3 (27.3) | 4.6 (26.4) | 12.7 (32.0) | 10.4 (20.2)
  Body Image: Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Body Image: Week 52 | 8.9 (20.2) | -5.0 (26.7) | 7.0 (31.3) | 9.6 (24.0)
  Fatigue: Week 12 | 10.049 (21.253) | 8.424 (19.509) | 6.250 (20.880) | 10.541 (22.488)
  Fatigue: Week 24: number analyzed (Participants) | 45 | 45 | 30 | 50
  Fatigue: Week 24 | 9.861 (23.175) | 10.972 (20.127) | 6.458 (17.790) | 10.625 (23.257)
  Fatigue: Week 36: number analyzed (Participants) | 41 | 40 | 27 | 44
  Fatigue: Week 36 | 9.909 (19.664) | 9.219 (20.363) | 7.407 (17.076) | 15.057 (28.220)
  Fatigue: Week 44: number analyzed (Participants) | 36 | 36 | 28 | 36
  Fatigue: Week 44 | 10.764 (17.205) | 12.153 (18.717) | 9.821 (16.876) | 12.500 (22.952)
  Fatigue: Week 52: number analyzed (Participants) | 31 | 36 | 27 | 35
  Fatigue: Week 52 | 12.500 (22.765) | 9.722 (20.291) | 9.954 (18.036) | 9.464 (21.404)

24. Secondary Outcome: Change From Baseline in Patient Global Assessment Score (PtGA) at Weeks 12, 24, 36, 44, and 52
Description: The PtGA assesses disease activity on a 10 cm numeric rating scale (NRS; 0 to 10 cm). The scale for the assessment ranges from "very well" (0) to "very poor" (10).
Time Frame: Week 12, 24, 36, 44, and 52
Population: The FAS included all randomized participants. Only participants with observed data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 51 | 44 | 31 | 65
Score on a scale
  Week 12 | -0.9 (2.8) | -1.1 (1.9) | -1.8 (3.0) | -1.7 (2.2)
  Week 24: number analyzed (Participants) | 45 | 44 | 30 | 49
  Week 24 | -1.9 (2.6) | -1.2 (2.7) | -1.7 (2.7) | -2.2 (2.1)
  Week 36: number analyzed (Participants) | 40 | 37 | 28 | 44
  Week 36 | -2.0 (2.6) | -1.7 (2.5) | -1.6 (2.3) | -2.6 (2.6)
  Week 44: number analyzed (Participants) | 36 | 35 | 28 | 36
  Week 44 | -2.1 (3.0) | -2.1 (2.8) | -2.0 (2.8) | -2.6 (2.3)
  Week 52: number analyzed (Participants) | 30 | 33 | 27 | 35
  Week 52 | -2.3 (2.7) | -1.8 (2.5) | -2.6 (2.5) | -2.1 (2.8)

25. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any negative medical occurrence linked to an intervention in humans, regardless of its relation to the intervention. Treatment-emergent AEs (TEAEs) were those that occurred after the first intervention dose. A serious adverse event (SAE) included outcomes such as death, life-threatening situations, hospitalization or an extended hospital stay, significant incapacity, congenital defects, or other crucial medical events. AE severity followed the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 scale: grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), and grade 5 (death). Clinically significant laboratory results or other assessments (e.g., ECGs, scans, vital signs) that worsened from baseline and were deemed important by the investigator, independent of disease progression, were also considered.
Time Frame: Up to approximately 68 weeks
Population: The Safety Analysis Set (SAS) included all randomized participants who received at least 1 dose of investigational product (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 62 | 58 | 36 | 87
Participants
  All TEAEs | 42 | 47 | 23 | 71
  Fatal AEs | 0 | 0 | 0 | 0
  SAEs | 6 | 7 | 5 | 3

26. Secondary Outcome: Serum Concentration of Rozibafusp Alfa
Time Frame: Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 36, Week 44, Week 52, Week 56, Week 60, Week 64, and Week 68
Population: The pharmacokinetic (PK) concentration analysis set contained all participants who received at least one dose of IP and had at least one quantifiable PK sample collected. PK concentration data was analyzed according to the actual treatment received.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 0 | 57 | 36 | 84
μg/mL
  Week 1 |  | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 4: number analyzed (Participants) | 0 | 49 | 31 | 68
  Week 4 |  | 1.29 (1.34) | 20.7 (10.8) | 26.2 (17.1)
  Week 8: number analyzed (Participants) | 0 | 46 | 29 | 61
  Week 8 |  | 1.70 (1.93) | 26.6 (15.7) | 40.7 (21.8)
  Week 12: number analyzed (Participants) | 0 | 42 | 23 | 66
  Week 12 |  | 2.05 (2.03) | 31.3 (16.5) | 46.8 (24.6)
  Week 16: number analyzed (Participants) | 0 | 40 | 24 | 62
  Week 16 |  | 2.58 (2.67) | 29.8 (18.9) | 47.0 (28.4)
  Week 20: number analyzed (Participants) | 0 | 40 | 26 | 55
  Week 20 |  | 3.42 (3.15) | 35.4 (19.8) | 48.9 (30.0)
  Week 24: number analyzed (Participants) | 0 | 41 | 27 | 53
  Week 24 |  | 3.69 (3.37) | 35.8 (19.1) | 55.5 (30.6)
  Week 36: number analyzed (Participants) | 0 | 36 | 25 | 43
  Week 36 |  | 3.62 (3.73) | 40.5 (20.7) | 54.7 (35.9)
  Week 44: number analyzed (Participants) | 0 | 38 | 24 | 38
  Week 44 |  | 2.98 (3.78) | 39.0 (18.6) | 54.1 (38.3)
  Week 52: number analyzed (Participants) | 0 | 35 | 23 | 32
  Week 52 |  | 4.15 (4.50) | 43.8 (25.3) | 51.6 (30.8)
  Week 56: number analyzed (Participants) | 0 | 33 | 18 | 34
  Week 56 |  | 0.230 (0.495) | 11.3 (8.03) | 13.3 (12.4)
  Week 60: number analyzed (Participants) | 0 | 29 | 20 | 34
  Week 60 |  | 0.00346 (0.0120) | 3.45 (4.31) | 3.08 (4.45)
  Week 64: number analyzed (Participants) | 0 | 35 | 23 | 36
  Week 64 |  | 0.0 (0.0) | 0.609 (1.07) | 0.718 (1.41)
  Week 68: number analyzed (Participants) | 0 | 39 | 22 | 36
  Week 68 |  | 0.0 (0.0) | 0.0484 (0.125) | 0.102 (0.271)

27. Secondary Outcome: Terminal Half-life of Rozibafusp Alfa
Time Frame: Up to Week 68
Population: Per the SAP, data for this outcome measure was not to be analyzed unless it could be adequately estimated.
Arm/Group | Placebo | Rozibafusp Alfa 70mg | Rozibafusp Alfa 280mg | Rozibafusp Alfa 420mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 68 weeks
Description: The SAS included all randomized participants who received at least 1 dose of IP. All-cause mortality is reported for all participants enrolled/randomized in the study. Treatment emergent serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Rozibafusp Alfa 70 mg: Participants received Rozibafusp Alfa 70mg SC Q2W for a maximum duration of 52 weeks.
- Rozibafusp Alfa 280 mg: Participants received Rozibafusp Alfa 280mg SC Q2W for a maximum duration of 52 weeks.
- Rozibafusp Alfa 420 mg: Participants received Rozibafusp Alfa 420mg SC Q2W for a maximum duration of 52 weeks.
Arm/Group | Placebo | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 280 mg | Rozibafusp Alfa 420 mg
All-Cause Mortality (participants affected / at risk) | 0/62 | 1/58 | 0/36 | 0/88
Serious Adverse Events (participants affected / at risk) | 6/62 | 7/58 | 5/36 | 3/87
Other Adverse Events (participants affected / at risk) | 29/62 | 34/58 | 20/36 | 51/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Rozibafusp Alfa 70 mg (N=58) | Rozibafusp Alfa 280 mg (N=36) | Rozibafusp Alfa 420 mg (N=87)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Serositis (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
SLE arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Rozibafusp Alfa 70 mg (N=58) | Rozibafusp Alfa 280 mg (N=36) | Rozibafusp Alfa 420 mg (N=87)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1 | 4
Injection site erythema (General disorders) | 2 | 0 | 3 | 1
Injection site reaction (General disorders) | 1 | 1 | 1 | 5
Oedema peripheral (General disorders) | 1 | 3 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 1 | 4
Bronchitis (Infections and infestations) | 3 | 2 | 2 | 4
COVID-19 (Infections and infestations) | 5 | 13 | 3 | 19
Influenza (Infections and infestations) | 1 | 3 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3 | 1 | 8
Upper respiratory tract infection (Infections and infestations) | 8 | 6 | 6 | 8
Urinary tract infection (Infections and infestations) | 6 | 9 | 4 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 5
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 5
Headache (Nervous system disorders) | 3 | 5 | 3 | 8
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Hypertension (Vascular disorders) | 1 | 3 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT04058028/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT04058028/SAP_001.pdf